CLINICAL TRIAL: NCT00878579
Title: A Study to Evaluate the Safety and Effectiveness of the PDS System to Treat Back Pain Associated With Degenerative Disc Disease
Brief Title: Percutaneous Dynamic Stabilization (PDS) System Versus Fusion for Treating Degenerative Disc Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Termination
Sponsor: Interventional Spine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDS-002-DDD
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Lumbar Degenerative Disc Disease
Keywords: back pain; Spine; Spinal; Lower back pain; Lumbar; Lumbar Pain; DDD; Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDS System (Experimental)
  Interventions: Device: PDS System
- Fusion (Active Comparator)
  Interventions: Device: Fusion

INTERVENTIONS:
Device: PDS System — Percutaneous Dynamic Stabilization System
  Arms: PDS System
Device: Fusion — Transforaminal Interbody Fusion (TLIF) with Autograft and Pedicle Screws
  Arms: Fusion

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the PDS System compared to the surgical control of posterolateral fusion with autograft and pedicle screw fixation for the treatment of one or two levels from L3-S1 to relieve back pain associated with degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of DDD (back pain with degeneration of the disc by patient history, physical exam, and radiographic studies and with one or more of the following factors:

   * Osteophyte formation of facet joints or vertebral endplates
   * Facet joint degeneration (no more than mild to moderate)
   * Subjects with ≤50% collapse of disc as compared to the adjacent level
   * Subjects with or without a contained herniated nucleus pulposus <5 mm and no free fragment
2. Skeletally mature subjects aged between 18 and 70 years of age inclusive.
3. Subjects with primarily back pain associated with degenerative disc disease of the lumbar spine at one level or two adjacent levels from L3 through S1. Subjects may have a lesser degree of leg pain at the same level(s).
4. Subjects who require surgical or minimally invasive intervention, who have failed to adequately improve following 6 months of non-operative therapy.
5. Subject is a surgical candidate for a posterior approach to the lumbar spine and is suitable for fusion using pedicle screw systems
6. Subjects with a minimum baseline Oswestry Score of 40% (20/50).
7. Subjects with a minimum baseline VAS Score of 40/100 mm.
8. MRI diagnostic for DDD within 3 months of the screening visit.
9. Subjects who are mentally, physically and psychosocially able to cooperate with the study procedures and return for all required follow-up visits.
10. Subjects who are able to understand this study and have given voluntary, written informed consent to participate in this study.

Exclusion Criteria:

1. Subjects who have leg pain greater than back pain.
2. Subjects with severe facet degeneration, radiographic findings of severe facet joint disease, degeneration or misshapen facet(s) or structural anomalies at the target level(s) that would preclude placement of the PDS device or pedicle screw systems.
3. Subjects who require a pedicle screw smaller than 4.5 mm.
4. Subjects with Modic 3 bone changes at the target level(s).
5. Spondylolisthesis > Grade 1 and/or spondylolysis at the target level(s).
6. Subjects with myelopathy or cauda equina syndrome, defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder dysfunction (retention or incontinence).
7. Subjects with fixed motor deficit and/or peripheral neuropathy.
8. Subjects with prior discectomy at the target level(s).
9. Subjects with prior spine surgery, trauma, metastatic disease, or spinal deformity due to scoliosis (Cobb angle > 15 degrees) or kyphosis (> 11 degrees) at any lumbar level.
10. Subjects who have used any investigational drug or device within the past 30 days or have had an experimental spinal implant at any time.
11. Subjects with active local or systemic infection.
12. Subjects with osteoporosis. A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen subjects. If DEXA is required, exclusion will be defined as a DEXA bone density measured T scored < -1.0.
13. Subjects with metabolic bone disease (e.g. osteomalacia, Paget's disease).
14. Subjects with rheumatoid arthritis or other autoimmune spondyloarthropathies.
15. Subjects with a systemic disease that compromises life expectancy (e.g. HIV, AIDS, hepatitis) or are on immuno-suppressive agents.
16. Subjects who are taking any drug known to potentially interfere with bony/soft tissue healing, (e.g., steroids at any dose daily within the last 12 months).
17. Subjects with active malignancy: A subject with a history of any invasive malignancy (except non-melanoma skin cancer), unless s/he has been treated with curative intent and there have been no clinical signs or symptoms of malignancy for at least 5 years.
18. Subjects with a known allergy to titanium and/or polycarbonate urethane (PCU).
19. Subjects who have existing conditions or pending litigation claims that could compromise their participation, follow-up care, or treatment outcomes (e.g., drug or alcohol abuse).
20. Subjects with a BMI of ≥ 40 kg/m2 or weight > 275 pounds (125 kg).
21. Subjects who are pregnant or are planning a pregnancy during the study period.
22. Subjects who are prisoners.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Improvement in Oswestry Disability Index (ODI) | 2 Years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati, Ohio
  - Willow Grove, Pennsylvania